CLINICAL TRIAL: NCT01227421
Title: A Randomized, Double-Blind, Placebo Controlled Study of Nitazoxanide in Adults and Adolescents With Acute Uncomplicated Influenza
Brief Title: Safety and Efficacy Study of Nitazoxanide in the Treatment of Acute Uncomplicated Influenza
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM08-3001
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Influenza
Keywords: influenza
MeSH Terms: conditions — Influenza, Human | interventions — nitazoxanide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nitazoxanide, Placebo (Active Comparator): 300 mg nitazoxanide tablet and 1 placebo tablet twice daily for 5 days
  Interventions: Drug: Nitazoxanide
- Nitazoxanide, Nitazoxanide (Active Comparator): Two 300 mg nitazoxanide tablets(600mg) twice daily for 5 days
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): 2 placebo tablets twice daily for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitazoxanide — Tablets, 300 mg (one 300 mg tablet + 1 placebo tablet) with food twice daily for 5 days
  Other Names: Alinia, NTZ
  Arms: Nitazoxanide, Placebo
Drug: Nitazoxanide — Tablets, 600 mg (two 300 mg tablets) with food twice daily for 5 days
  Other Names: Alinia, NTZ
  Arms: Nitazoxanide, Nitazoxanide
Drug: Placebo — Tablets, (2 tablets) twice daily with food for 5 days
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This is a randomized clinical trial designed to evaluate the safety/efficacy of two dosing regimens of oral nitazoxanide compared to placebo in the treatment of acute uncomplicated influenza in adults and adolescents. The investigators hypothesize that treatment with Nitazoxanide will reduce the duration of symptoms in patients with confirmed influenza infection. Secondarily, the investigators hypothesize that treatment with nitazoxanide will reduce the complications of influenza, severity of symptoms, time lost from work, time to return to normal daily activities.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo Controlled Study of Nitazoxanide in Adults and Adolescents with Acute Uncomplicated Influenza. The primary objectives of this study are to demonstrate the efficacy of nitazoxanide administered 300 mg two times per day for 5 days or 600 mg two times per day for 5 days in reducing the time to resolution of all clinical symptoms of influenza.

The study will also evaluate pharmacokinetics of nitazoxanide in a subset of 24 patients and the safety of the nitazoxanide regimen compared to a placebo via analysis of adverse events and laboratory safety tests.

Blood samples will be collected for all patients at baseline, day 7 and day 28, and for a subset of 24 patients aged 18-65 years (pharmacokinetics subset) on day 2. Urine samples will be collected at baseline and day 7. Nasal swabs will be collected at baseline and day 7 for all patients and on days 2, 3, 4 and 5 for a subset of patients (approximately 20% of patients).

ELIGIBILITY:
INCLUSION CRITERIA

* age 12 to 65 years
* Presence of clinical signs, respiratory symptoms and constitutional symptoms compatible with influenza infection:

  1. fever,
  2. at least one of the following respiratory symptoms: cough, sore throat, nasal discharge, nasal congestion, sneezing.
  3. At least one of the following constitutional symptoms: headache, myalgia, seats, chills, fatigue of any severity (mild, moderate, severe)
* Confirmation of Influenza A or B infection in the local community
* Onset of illness no more than 48 hours before presentation. Time of onset of illness is defined as either the earlier of (1) the time when the temperature was first measured as elevated, or (2) the time when the patient experienced the presence of at least one respiratory symptom AND the presence of at least one constitutional symptom.
* willing and able to comply with protocol requirements and provide informed consent

EXCLUSION CRITERIA:

* severity of illness requiring or anticipated to require in-hospital care
* High risk of complications from influenza as follows:

  1. persons with asthma or other chronic pulmonary diseases
  2. persons with hemodynamically significant cardiac disease
  3. persons who have immunosuppressive disorders or receiving immunosuppressive therapy
  4. persons infected with Human Immunodeficiency Virus (HIV)
  5. persons with sickle cell anemia or other hemoglobinopathies
  6. persons with diseases requiring long-term aspirin therapy
  7. persons with chronic renal dysfunction
  8. persons with liver disorders
  9. Persons with cancer
  10. Persons with chronic metabolic disease such as diabetes and inherited mitochondrial disorders
  11. Persons with neuromuscular disorders, seizure disorders, or cognitive dysfunction
  12. Residents of any age of nursing homes or long-term institutions.
* Females of child bearing age who are pregnant, breastfeeding or sexually active without birth control
* vaccination for influenza or H1N1 (Swine Flu) on or after August 1, 2010
* treatment with antiviral medication such as oseltamivir, zanamivir, amantadine, or rimantadine within 30 days of screening.
* Prior treatment with nitazoxanide within 30 days prior to screening.
* subjects with active respiratory allergies or expected to require anti-allergy medications during the study period.
* known sensitivity to nitazoxanide
* subjects unable to take oral medication
* subjects with chronic kidney or liver disease
* Presence of any other pre-existing chronic infection that is undergoing or requiring medical therapy

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rossignol, M.D., Ph.D., Study Director — Romark Laboratories L.C.
Locations (1):
- Health Sciences Research Center, Elmira, New York, United States

REFERENCES:
- [Derived] Haffizulla J, Hartman A, Hoppers M, Resnick H, Samudrala S, Ginocchio C, Bardin M, Rossignol JF; US Nitazoxanide Influenza Clinical Study Group. Effect of nitazoxanide in adults and adolescents with acute uncomplicated influenza: a double-blind, randomised, placebo-controlled, phase 2b/3 trial. Lancet Infect Dis. 2014 Jul;14(7):609-18. doi: 10.1016/S1473-3099(14)70717-0. Epub 2014 May 19. PMID 24852376

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitazoxanide 300mg: 300 mg nitazoxanide twice daily with food for 5 days
- Placebo: placebo tablet twice daily with food for 5 days
- Nitazoxanide 600mg: 2X 300 mg controlled release tablet twice daily with food for five days
Period: Overall Study
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Started | 201 | 212 | 211
Completed | 190 | 194 | 201
Not Completed | 11 | 18 | 10
Not completed — Lost to Follow-up | 6 | 7 | 5
Not completed — Adverse Event | 2 | 7 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Randomized in error | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg | Total
Number analyzed (Participants) | 201 | 212 | 211 | 624
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 21 | 20 | 66
  Between 18 and 65 years | 176 | 189 | 188 | 553
  >=65 years | 0 | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (12.6) | 31 (13.3) | 32 (13.2) | 31 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 122 | 129 | 355
  Male | 97 | 90 | 82 | 269
Region of Enrollment [Number; unit: participants]
  United States | 201 | 212 | 211 | 624

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of All Clinical Symptoms of Influenza as Reported by the Subjects
Description: The primary efficacy analysis for this study was to demonstrate the efficacy of Nitazoxanide (NTZ) administered as 300 mg b.i.d. for 5 days or 600 mg b.i.d. for 5 days in reducing the time to resolution of all clinical symptoms of influenza in patients with laboratory confirmed influenza infection
Time Frame: Up to 28 days
Population: 624 patients were enrolled based on inclusion/exclusion criteria. The primary efficacy analysis was conducted on the 257 patients with laboratory confirmed influenza.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 89 | 89 | 79
Hours | 109.1 [81.5 to 151.9] | 116.7 [91.3 to 144.0] | 95.5 [71.2 to 125.8]

2. Secondary Outcome: Time to Resolution of Each Individual Symptom of Influenza as Reported by the Subjects
Description: Time in hours (Median and Interquartile range)
Time Frame: at least 28 days
Population: 624 patients were enrolled based on inclusion/exclusion criteria. Secondary efficacy analyses were conducted on the 257 patients with laboratory confirmed influenza.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 89 | 89 | 79
Hours
  Nasal Congestion | 84 [72 to 92] | 81 [67 to 92] | 60 [48 to 74]
  Runny Nose | 48 [37 to 82] | 42 [36 to 56] | 43 [36 to 51]
  Sore Throat | 63 [48 to 74] | 52 [36 to 72] | 50 [31 to 60]
  Cough | 96 [75 to 117] | 104 [84 to 111] | 84 [60 to 105]
  Headache | 42 [36 to 60] | 48 [39 to 60] | 39 [30 to 49]
  Myalgia | 46 [36 to 52] | 46 [39 to 57] | 42 [30 to 51]
  Fatigue | 65 [52 to 83] | 69 [60 to 72] | 60 [38 to 69]
  Sweats / Chills | 36 [34 to 42] | 36 [27 to 42] | 36 [26 to 42]
  Fever | 36 [28 to 41] | 31 [24 to 41] | 36 [24 to 42]

3. Secondary Outcome: Mean Change (Standard Deviation)in 50% Tissue Culture Infective Dose (TCID50) Viral Titer From Baseline
Description: Change in viral titer presented as logarithm with base 10 (log10) 50% Tissue Culture Infective Dose (TCID50)
Time Frame: 7 days
Population: Analysis conducted on 113 patients from intensive virologic follow up group with laboratory confirmed influenza
Measure: Mean (Standard Deviation); unit: LOG10 Titer
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 33 | 41 | 39
LOG10 Titer
  Day 2 | -0.58 (1.4) | -0.03 (1.7) | -1.11 (1.7)
  Day 3 | -1.26 (1.8) | -1.21 (2.2) | -1.84 (1.7)
  Day 4 | -1.86 (1.9) | -1.65 (1.9) | -2.58 (1.3)
  Day 5 | -2.46 (1.8) | -2.41 (1.8) | -2.55 (1.4)
  Day 7 | -2.82 (1.6) | -2.79 (1.8) | -3.01 (1.4)

4. Secondary Outcome: Mean Change in RT-PCR (Reverse Transcription Polymerase Chain Reaction) Viral Titer From Baseline
Description: Change in viral titer logarithm with base 10 (log10) Ribonucleic Acid (RNA)copies
Time Frame: 7 days
Population: Analysis conducted on 113 patients from the intensive virologic follow up group with laboratory confirmed influenza
Measure: Mean (Standard Deviation); unit: LOG10 RNA copies
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 33 | 41 | 39
LOG10 RNA copies
  Day 2 | -0.63 (1.4) | -0.22 (1.7) | -0.73 (1.5)
  Day 3 | -1.34 (1.4) | -0.92 (2.0) | -1.64 (1.7)
  Day 4 | -1.75 (1.5) | -1.63 (1.8) | -2.21 (1.4)
  Day 5 | -2.42 (1.5) | -2.49 (1.7) | -2.44 (1.4)
  Day 7 | -2.97 (1.3) | -2.82 (1.6) | -3.08 (1.3)

5. Secondary Outcome: Time to Cessation of Viral Shedding Measure by 50% Tissue Culture Infective Dose (TCID50)
Description: Median time in hours
Time Frame: 28 days
Population: Analysis performed on 107 patients from the intensive virologic follow up population with laboratory confirmed influenza
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 31 | 39 | 37
Hours | 77.0 [46 to 141] | 91.3 [48 to 143] | 71.8 [38 to 142]

6. Secondary Outcome: Time to Return to Normal Daily Activities
Description: Time in hours as reported by patient
Time Frame: 28 days
Population: Analysis conducted on 257 patients with laboratory confirmed influenza
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 89 | 89 | 79
Hours | 84.2 [49 to 117] | 82.1 [59 to 115] | 84.0 [60 to 115]

7. Secondary Outcome: Symptom Severity Score Hours
Description: Sum of the symptom severity score hours from first dose to resolution of symptoms. Patients rated each symptom's severity on a score from 0 to 3 (0=absent, 1=mild, 2=moderate, 3=severe). Total symptom severity score hours were calculated by multiplying the sum of the severity scores by duration of symptoms.
Time Frame: 28 days
Population: Analysis conducted for 257 patients with laboratory confirmed influenza
Measure: Mean (Standard Deviation); unit: symptom score *hour
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 89 | 89 | 79
symptom score *hour | 1035.1 (765) | 1220.9 (592) | 1125.2 (681)

8. Secondary Outcome: Time Loss From Work
Description: Time loss from work
Time Frame: 28 days
Population: Analysis conducted on 241 patients with laboratory confirmed influenza excluding those who are unemployed
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 84 | 82 | 75
days | 2.6 [2.17 to 3.11] | 3.0 [2.43 to 3.49] | 3.3 [2.75 to 3.92]

9. Secondary Outcome: Complications of Influenza
Description: Proportion of patients with a complication of influenza during the course of the study
Time Frame: 28 days
Population: All patients who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 201 | 212 | 211
Participants
  Bronchitis | 10 | 3 | 7
  Sinusitis | 6 | 6 | 2
  Pneumonia | 1 | 2 | 1
  Pleurisy | 0 | 1 | 0
  Otitis | 3 | 3 | 1

10. Secondary Outcome: Influenza Antibody Response Titer Change: Influenza A 2009 H1N1
Description: change in influenza antibody titer for Influenza A 2009 H1N1
Time Frame: 28 days
Population: Member of the intensive virologic follow up group with laboratory confirmed Influenza A 2009 H1N1
Measure: Median (Inter-Quartile Range); unit: Fold change in antibody titer
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 26 | 34 | 36
Fold change in antibody titer | 2 [1 to 8] | 2 [1 to 5] | 2 [1 to 4]

11. Secondary Outcome: Influenza Antibody Response: Influenza A H3N2
Description: Change in antibody titer for Influenza A H3N2
Time Frame: 28 days
Population: Members of the intensive virologic follow up group with laboratory confirmed influenza A H3N2
Measure: Median (Inter-Quartile Range); unit: Fold change in antibody titer
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 15 | 16 | 12
Fold change in antibody titer | 8 [4 to 16] | 16 [2 to 56] | 16 [10 to 30]

12. Secondary Outcome: Influenza Antibody Response: Influenza B
Description: Change in antibody titer for Influenza B
Time Frame: 28 days
Population: Members of intensive virologic follow up group with laboratory confirmed Influenza B
Measure: Median (Inter-Quartile Range); unit: Fold change in antibody titer
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 21 | 20 | 17
Fold change in antibody titer | 4 [1 to 8] | 3 [1 to 4] | 4 [1 to 10]

13. Secondary Outcome: Influenza Antibody Response: Seroprotection and Seroconversion for Patients With Influenza A 2009 H1N1
Description: Proportion of patients seroprotected or seroconverted at day 28
Time Frame: 28 days
Population: Members of intensive virologic follow up group with laboratory confirmed Influenza A 2009 H1N1
Measure: Number; unit: Participants
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 26 | 34 | 36
Participants
  Seroprotected at day 28 | 11 | 14 | 12
  Seroconverted at day 28 | 11 | 12 | 11

14. Secondary Outcome: Influenza Antibody Response: Seroprotection and Seroconversion for Patients With Influenza A H3N2
Description: Proportion of patients seroprotected and seroconverted at day 28
Time Frame: 28 days
Population: Members of intensive virologic follow up group with laboratory confirmed Influenza A H3N2
Measure: Number; unit: Participants
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 15 | 16 | 12
Participants
  Seroprotected at day 28 | 14 | 12 | 12
  Seroconverted at day 28 | 13 | 12 | 12

15. Secondary Outcome: Influenza Antibody Response: Seroprotection and Seroconversion for Influenza B
Description: Proportion of patients seroprotected and seroconverted at day 28
Time Frame: 28 days
Population: Members of intensive virologic follow up group with laboratory confirmed Influenza B
Measure: Number; unit: Participants
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Number analyzed (Participants) | 21 | 20 | 17
Participants
  Seroprotected at day 28 | 14 | 13 | 13
  Seroconverted at day 28 | 12 | 10 | 13

ADVERSE EVENTS:
Arm/Group | Nitazoxanide 300mg | Placebo | Nitazoxanide 600mg
Serious Adverse Events (participants affected / at risk) | 0/201 | 1/212 | 1/211
Other Adverse Events (participants affected / at risk) | 10/201 | 7/212 | 25/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide 300mg (N=201) | Placebo (N=212) | Nitazoxanide 600mg (N=211)
moderate pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Patient experienced influenza symptoms 18 hours prior to 600mg NTZ enrollment. Patient had Body Mass Index (BMI) 48.5, history of osteoarthritis & hypertension. Tests reveal 2009 H1N1. Investigator noted adverse event was not related to study drug.
respiratory syncytial virus type A (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Patient presented influenza type symptoms 44 hours prior to enrollment to placebo group. Completed medication & symptoms resolved. Day 17, admitted to hospital with hypertensive emergency. Investigator noted adverse event not related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide 300mg (N=201) | Placebo (N=212) | Nitazoxanide 600mg (N=211)
Chromaturia (Renal and urinary disorders) | 6 (6) | 0 (0) | 8 (8)
Mild Diarrhea (Gastrointestinal disorders) | 4 (4) | 7 (7) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Presentation and/or publication is encouraged provided the Sponsor is notified in advance and given the opportunity to review the manuscript or abstract 30 days prior to its submission for presentation at a scientific meeting or for publication in a scientific journal. The investigators will have complete autonomy regarding the content and wording including the decision of whether or not to publish.